CLINICAL TRIAL: NCT07324798
Title: Prospective Study of siMultaneous Adaptive RadioTherapy for Local Boost for Prostate and Bladder Cancers (SMART-B01)
Brief Title: Adaptive Radiotherapy for Genitourinary Cancers
Acronym: SMART-B01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NINGNING LU, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-020503
Record Dates: First submitted 2025-12-02; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer (Post Prostatectomy); Bladder Cancer
Keywords: prostate cancer; bladder cancer; adaptive radiotherapy; post-prostatectomy; bladder-conserving treatment
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Pts will receive adaptive boost for clinically significant disease
  Interventions: Radiation: adaptive RT

INTERVENTIONS:
Radiation: adaptive RT — Prostate cancer pts post-prostatectomy：95%PTVboost 7Gy/3.5Gy/2f，95%PTV 66Gy/2.0Gy/33f，w/o 95%PTVp 50Gy/2.0Gy/25f Bladder cancer pts with bladder-conserving txt：95%PGTV 18Gy/6.0Gy/3f，95%PTV 50Gy/2.0Gy/25f，w/o 95%PTVp 50Gy/2.0Gy/25f

SUMMARY:
The goal of this clinical trial is to learn if adaptive radiation boost works to treat genitourinary cancers, esp. in the context of prostate cancer patients with post-prostatectomy local relapse and bladder cancer patients with bladder-conserving treatment. It will also learn about the safety and efficacy of adaptive boost. The main questions it aims to answer are:

Does adaptive boost lower the toxicities? Does adaptive boost maintain or improve the clinical efficacy?

Participants will:

Undergo adaptive boost on 1.5-Tesla MR-Linac Visit the clinic once every 2 weeks during RT, and every 3 months post-ART Keep a regular QOL questinnaire completion

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed or metastatic/recurrent pathologically confirmed urological tumors, clinically assessed as suitable for adaptive radiotherapy;
* Age ≥ 18 years;
* ECOG performance status score 0-2;
* No prior radiotherapy history within the current radiation field;
* No contraindications for MRI scanning;
* No contraindications for radiotherapy.

Exclusion Criteria:

* Patients with contraindications to radiotherapy;
* Patients unable to tolerate MRI or with contraindications to MRI scanning.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute GU and GI toxicities as per NCI-CTC 5.0 criteria 3-months post RT | 3-months post-RT

SECONDARY OUTCOMES:
Quality-of-Life, general | Baseline, 1-month post-RT, every 3 months till 2-years post-RT
  general quality-of-life questionaaires as per EORTC QLQ-C30
Local control | 2-year
  local control
disease-free survival | 2-year
  disease-free survival
Late toxicities | 2-year
  Late GU and GI toxicities as per RTOG scales
Quality-of-Life, GU (genitourinary) and GI (gastrointestinal) scales | Baseline, 1-month post-RT, every 3 months till 2-years post-RT
  GU quality-of-life questionaaires as per EORTC QLQ-NMIBC24
Quality-of-Life, GU (genitourinary) and GI (gastrointestinal) scales | Baseline, 1-month post-RT, every 3 months till 2-years post-RT
  quality-of-life questionaaires as per EORTC QLQ- BLM30
Quality-of-Life, GU (genitourinary) and GI (gastrointestinal) scales | Baseline, 1-month post-RT, every 3 months till 2-years post-RT
  quality-of-life questionaaires as per BCI
Quality-of-Life, GU (genitourinary) and GI (gastrointestinal) scales | Baseline, 1-month post-RT, every 3 months till 2-years post-RT
  quality-of-life questionaaires as per FACT-BL
Quality-of-Life, GU (genitourinary) and GI (gastrointestinal) scales | Baseline, 1-month post-RT, every 3 months till 2-years post-RT
  quality-of-life questionaaires as per FACT-P
Quality-of-Life, GU (genitourinary) and GI (gastrointestinal) scales | Baseline, 1-month post-RT, every 3 months till 2-years post-RT
  quality-of-life questionaaires as per EPIC-26
Quality-of-Life, sexual scales | Baseline, 1-month post-RT, every 3 months till 2-years post-RT
  quality-of-life questionaaires as per IIEF-5

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, National Cancer Center, CAMS & PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided